CLINICAL TRIAL: NCT02863939
Title: Quantitation of Cardiac Output Change by Impedance Cardiography in Subjects Undergoing Exercise Gated Stress/Rest Tc-99m CZT-SPECT MPI
Acronym: NICAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NICAS 1.0
Record Dates: First submitted 2016-07-24; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NICAS (Other): There is only one arm - a single cohort. All patients undergoing the nuclear stress test will also have the NICAS evaluation.
  Interventions: Device: Single photon emission computed tomography myocardial perfusion imaging; Other: exercise

INTERVENTIONS:
Device: Single photon emission computed tomography myocardial perfusion imaging — a novel cadmium-zinc-telluride (CZT) SPECT camera
Other: exercise

SUMMARY:
The aim of this study is to test for an early post-stress cardiac output (CO) change by impedance cardiography and its relation to the severity and extent of myocardial ischemia and angiographic coronary disease in subjects undergoing exercise stress testing using a novel cadmium-zinc-telluride (CZT) SPECT camera.

DETAILED DESCRIPTION:
Single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI) is a well-established noninvasive procedure for the evaluation and risk stratification of patients with coronary artery disease (CAD) (1). However, it has been recognized that in certain patients SPECT MPI is unable to detect the presence of or underestimates the extent of CAD. The fact that moderate to severe perfusion defects are noted in less than half of the patients with significant left main disease (2) has stimulated studies to improve the diagnostic accuracy of SPECT MPI. Such studies have analyzed post-stress parameters such as left ventricular (LV) ejection fraction (EF) (3, 4), wall motion abnormalities (5) and transient LV dilation (6) with images acquired on conventional Anger cameras as long as 60 minutes after the stress tracer injection. Such delayed assessment may miss early ischemic stunning as a result of its transient nature. However, detection of an early post-stress decrease in cardiac output (CO) may serve as a potential marker for the presence of significant or extensive ischemia. The aim of this study is to test for an early post-stress CO change by impedance cardiography and its relation to the severity and extent of myocardial ischemia and angiographic coronary disease in subjects undergoing exercise stress testing using a novel cadmium-zinc-telluride (CZT) SPECT camera.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Nuclear Cardiology Center for a clinically indicated exercise stress MPI study

Exclusion Criteria:

* known standard contraindications for ergometry
* anemia
* hyperthyroidism
* intra- and extra-cardiac shunts
* significant arrhythmia
* hemodialysis

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Ischemia | 15-20 minutes after stress test
  Inducible and reversible perfusion defects, representing myocardial ischemia
Cardiac Output | 15-20 minutes after exercise test
  Noninvasive evaluation of cardiac output using a novel algorithm based on impedenace